CLINICAL TRIAL: NCT03591991
Title: Effectiveness of Empagliflozin on Cardiac-renal Injury in Patients With Acute ST-segment-elevation Myocardial Infarction After Primary Percutaneous Coronary Intervention.
Brief Title: Empagliflozin on Cardiac-renal Injury in Patients With STEAMI Patients After Primary PCI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Dandan Li, Principal Investigator, Chinese PLA General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2018-04
Record Dates: First submitted 2018-07-08; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Reperfusion Injury, Myocardial
Keywords: Empagliflozin; Percutaneous coronary intervention; Reperfusion Injury; Microvascular protection; CI-AKI; No-Reflow Phenomenon
MeSH Terms: conditions — Myocardial Reperfusion Injury; Reperfusion Injury; No-Reflow Phenomenon | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Active Comparator): Patients will be randomized into two groups after enrolled. In Empagliflozin Group, the treatment started 30 minutes before PCI with a dose of 10 mg empagliflozin .After admission, patients were treated with 10 mg empagliflozin once daily for 3 mouths. The procedure will double blind to patients and investigators.
  Interventions: Drug: Empagliflozin
- Placebo group (Placebo Comparator): Patients will be randomized into two groups after enrolled. In Placebo Group, the treatment started 30 minutes before PCI with a dose of 10 mg Placebo .After admission, patients were treated with 10 mg Placebo once daily for 3 mouths. The procedure will double blind to patients and investigators.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Empagliflozin — After randomization,the treatment started 30 minutes before PCI with a dose of 10 mg empagliflozin . After admission, patients were treated with 10 mg empagliflozin once daily for 3 mouths.
  Arms: treatment group
Other: placebo — After randomization,the treatment started 30 minutes before PCI with a dose of 10 mg placebo . After admission, patients were treated with 10 mg placebo once daily for 3 mouths.
  Arms: Placebo group

SUMMARY:
This study is a single-center, prospective controlled trial addressing effectiveness of empagliflozin on cardiac-renal injury in patients with STEMI. Patients were randomized using a computer-generated sequence to either placebo or empagliflozin at a 1:1 ratio. Investigators, participants, and other study personnel were blinded to the assigned treatment for the duration of the study. The primary objective of this study is to investigate the effects of empagliflozin on myocardial infarct size measured using cardiac magnetic resonance (CMR) methods at 3 months. Key secondary endpoint: incidence of CIAKI within 48h after PCI. Inclusion Criteria:Patients with STEMI who were admitted to the Chinese PLA General Hospital were recruited between Ocotor 2018 and January 2019. STEMI was defined as typical chest pain lasting >30 minutes within the previous 12 hours, a clear ST-segment elevation of >0.1 mV in two or more contiguous electrocardiographic leads, and elevated blood levels of troponin T.Exclusion Criteria:Cardiogenic shock ,Hypoglycaemia ,Diabetic ketoacidosis,Genital and urinary infections,History of myocardial infarction,Stent thrombosis,Previous coronary artery bypass surgery,Type 1 Diabetes,Severe hepatic insufficiency,Advanced cancer patients,eGFR<30 ml/min.

All patients were informed of the potential risks (genital mycotic infections, urinary tract infections, diabetic ketoacidosis) associated with empagliflozin and then required to submit written informed consent before being included in the study. Patients were randomized using a computer-generated sequence to either placebo or empagliflozin at a 1:1 ratio. Patients in the empagliflozin group were treated with empagliflozin whereas patients in the control group were given placebo. The treatment started 30 minutes before PCI with a dose of 10 mg empagliflozin or placebo administered in the ambulance. After admission, patients were treated with 10 mg empagliflozin once daily for 3 mouths.

ELIGIBILITY:
Inclusion Criteria:

* Patients with STEMI who were admitted to the Chinese PLA General Hospital were recruited between June 2018 and September 2018.

Exclusion Criteria:

* Cardiogenic shock
* Hypoglycaemia
* Diabetic ketoacidosis
* Genital and urinary infections
* History of myocardial infarction
* Stent thrombosis
* Previous coronary artery bypass surgery
* Type 1 Diabetes
* Severe hepatic insufficiency
* Advanced cancer patients
* eGFR<30 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2018-10-01 (Estimated); Primary Completion 2019-01-31 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
final infarct size | 3 months after PCI
  the final infarct size measured by Cardiac magnetic resonance

SECONDARY OUTCOMES:
contrast induced acute kidney injury (CIAKI) | within 48 hours after PCI
  incidence of CIAKI within 48 hours after PCI